CLINICAL TRIAL: NCT06427096
Title: Effect of Healthy Family Program on Population Blood Pressure: A 1:1 Parallel Design, Multi-Center Cluster Randomized Trial
Brief Title: Effect of Healthy Family Program on Population Blood Pressure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Heart Health Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HFP2024
Record Dates: First submitted 2024-05-18; First posted 2024-05-23 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-06

CONDITIONS: Blood Pressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multifaceted intervention (Experimental): Residents in this group will receive multifaceted intervention including education for a healthy lifestyle, free provision of sodium substitute, weight management, physical exercise, BP monitoring, and appropriate antihypertensive treatment for individuals with hypertension.
  Interventions: Behavioral: Multifaceted intervention
- Usual care (No Intervention): Residents in this group will receive usual lifestyle and health care management.

INTERVENTIONS:
Behavioral: Multifaceted intervention — The multifaceted interventions is comprised of the following components:
  1. To establish a BP management team led by family health instructor. The team members also include family leaders and village doctors.
  2. To conduct multifaceted intervention, which includes education for a healthy lifestyle, free provision of sodium substitute, weight management, physical exercise, BP monitoring, and appropriate antihypertensive treatment for individuals with hypertension.
  Arms: Multifaceted intervention

SUMMARY:
This is a 1:1 parallel design, multi-center, cluster-randomized control trial. A total of 80 villages in Ruyang County, Henan Province, China, will be randomly assigned to the intervention group or control group. At least 100 participants from 30-50 families in each village will be included in this study. The intervention group will engage in a variety of strategies, including educating a healthy lifestyle, adopting a low-sodium diet, managing weight, participating in physical exercise, monitoring blood pressure, and undergoing antihypertensive treatment. These efforts will be led by family health instructors from the community. The control group will receive usual care. The primary endpoint of this study is the change of systolic blood pressure from baseline to 6 months, reported as the difference between intervention and control group.

DETAILED DESCRIPTION:
This cluster-randomized control trial aims to randomly allocate 80 villages in Ruyan County to either receive a multifaceted intervention led by family health instructors or continue with usual care. Each village will recruit around 100 individuals aged 40-80 years, with or without hypertension. In intervention villages, a blood pressure management team, headed by family health instructors and family leaders, will implement various strategies including promoting a low-sodium diet, weight management, physical exercise, blood pressure monitoring, and administering antihypertensive treatment. The intervention will span 6 months, followed by another 6-month follow-up period. The primary hypothesis posits that the mean systolic blood pressure change from baseline to 6 months will be higher in the intervention group compared to the control group. The objective of this "Health Family Program" is to evaluate the efficacy of a non-healthcare provider-led multifaceted intervention in enhancing healthy lifestyles and managing blood pressure among rural residents, regardless of their hypertension status, in China.

ELIGIBILITY:
1. Village screening:

   The suitable villages were initially screened according to the statistical information of the number of villages and households in Ruyang County.
2. Inclusion and Exclusion Criteria for the Family

Inclusion Criteria:

1. At least 2 participants between the age of 40-80 years meet the inclusion and exclusion criteria of family members and willing to participate in this study;
2. At least one family member can use the smartphone to upload BP values.

Exclusion Criteria:

1. Any family member participated in the other hypertension-related programs;
2. Inappropriate for the study decided by the healthy family instructor.

3.Inclusion and Exclusion Criteria for the Family Member

Inclusion Criteria:

1. 40-80 years old, regardless of BP level and antihypertensive treatment;
2. No travel plan for more than 1 month during the study period;
3. Written or fingerprinted informed consent form.

Exclusion Criteria:

1. Significant cognitive dysfunction;
2. With advanced tumor, dialysis, or other serious diseases;
3. Lying in bed for a long time or unable to take care of themselves;
4. Diagnosed of secondary hypertension;
5. Having birth plans in the next six months, pregnant or lactating women;
6. Other ineligible circumstances judged by the investigators.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8000 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2025-02-12 (Actual); Study Completion 2025-12-27 (Estimated)

PRIMARY OUTCOMES:
The changes of systolic blood pressure from baseline to 6 months | 6 months
  The systolic blood pressure changes from baseline to 6 months for all villagers, reported as the difference between intervention and control group.

SECONDARY OUTCOMES:
The changes of systolic blood pressure from baseline to 12 months | 12 months
  The systolic blood pressure changes from baseline to 12 months, reported as the difference between intervention and control group.
The changes of diastolic blood pressure from baseline to 6 months | 6 months
  The diastolic blood pressure changes from baseline to 6 months, reported as the difference between intervention and control group.
The proportion of participants with SBP≥130 or DBP≥80 mmHg at 6 months | 6 months
  The proportion of participants with SBP≥130 or DBP≥80 mmHg at 6 months
The proportion of participants with antihypertensive therapy at 6 months | 6 months
  The proportion of participants with antihypertensive therapy at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jun Cai, MD, Principal Investigator — Beijing Anzhen Hospital; Xin Du, MD, Principal Investigator — Beijing Anzhen Hospital; Craig S Anderson, MD, Principal Investigator — Institute of Science and Technology for Brain-Inspired Intelligence; Chao Jiang, MD, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Ruyang County People's Hospital, Luoyang, Henan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tang Y, Jiang C, Guo J, Li Y, Wang C, Chu SH, Wang Z, Wu Y, Hua C, Lu Y, Zhang S, Song Y, Han R, Dong J, Ma C, Cai J, Anderson CS, Du X. Study protocol for the healthy family program on population blood pressure: A multicenter, parallel group, cluster randomized, controlled trial in rural China. Am Heart J. 2025 May;283:70-80. doi: 10.1016/j.ahj.2025.01.014. Epub 2025 Jan 28. PMID 39884452